CLINICAL TRIAL: NCT02811549
Title: Benefits of the HiResolution Bionic Ear System in Adults With Asymmetric Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR0314
Record Dates: First submitted 2016-06-07; First posted 2016-06-23 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Hearing Loss; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases; Asymmetrical Hearing Loss; Single-Sided Deafness
Keywords: Cochlear Implant; HiRes™ 90K Advantage Implant; HiFocus™ Mid-Scala electrode; HiFocus™ 1J electrode; HiFocus Helix™ electrode; Cochlear Implantation; Listening Benefits; Adults; Cochlear Implant Benefit; Electrical Stimulation; HiRes™ Ultra Implant with HiFocus™ Mid-Scala electrode
MeSH Terms: conditions — Hearing Loss; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HiResolution Bionic Cochlear Implant (Experimental): HiRes 90K™ Advantage implant with HiFocus™ 1J electrode, HiRes 90K™ Advantage implant with the HiFocus Helix™ electrode, HiRes 90K™ Advantage implant with the HiFocus™ Mid-Scala electrode or the HiRes™ Ultra Implant with the HiFocus™ Mid-Scala electrode will be implanted in adults who have severe to profound sensorineural hearing loss in one ear, and up to moderate sensorineural hearing loss in the other ear (asymmetric hearing loss).
  Interventions: Device: HiResolution Bionic Cochlear Implant

INTERVENTIONS:
Device: HiResolution Bionic Cochlear Implant — HiRes 90K™ Advantage implant with HiFocus™ 1J electrode, HiRes 90K™ Advantage implant with the HiFocus Helix™ electrode, HiRes 90K™ Advantage implant with the HiFocus™ Mid-Scala electrode or the HiRes™ Ultra Implant with the HiFocus™ Mid-Scala electrode will be implanted in adults with eligible hearing profile.

SUMMARY:
The purpose of this feasibility study is to evaluate the benefit of unilateral implantation in adults who have severe to profound sensorineural hearing loss in one ear, and up to moderate sensorineural hearing loss in the other ear (asymmetric hearing loss).

ELIGIBILITY:
Inclusion Criteria:

General Requirements:

* Ability to provide Informed Consent
* 18 years of age or older
* English language proficiency
* Willingness to participate in all scheduled procedures outlined in the study investigational plan
* Willingness to use an approved cochlear implant signal processing strategy in an everyday listening program during study

Ear to be Implanted:

* Severe-to-profound sensorineural hearing loss (> 70 dB HL) as defined by the pure tone average for 500, 1000, 2000 and 4000 Hz
* CNC word recognition score ≤30% (tested in subject's everyday listening condition for that ear)
* Duration of severe-to-profound sensorineural hearing loss (≥ 70 dB HL) >3 months and ≤10 years in the ear to be implanted only

Contralateral (non-implanted) ear:

* Up to a moderate sensorineural hearing loss (<70 dB HL) as defined by the pure tone average for 500, 1000, 2000 and 4000 Hz
* CNC word recognition score >30% (tested in subject's everyday listening condition for that ear)

Exclusion Criteria:

* Previous experience with a cochlear implant
* Cochlear malformation or obstruction (i.e. ossification) that would preclude full insertion of electrode array in the ear to be implanted
* Medical or psychological conditions that contraindicate surgery or impact the ability to manage an implanted device or the study related procedures as determined by the investigator
* Diagnosis of auditory neuropathy/dys-synchrony in either the ear to be implanted or the contralateral ear
* Active middle-ear disease/infection in the ear to be implanted
* Unrealistic expectations regarding potential benefits, risks and limitations inherent to implant surgical procedures as determined by the investigator
* Unwillingness or inability of subject to comply with all investigational requirements as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Silverstein Institute, Sarasota, Florida
  - Virginia Mason Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators recruited study subjects from their clinical practices. The first patient first visit occurred on November 7, 2016 and last patient last visit occurred on March 25, 2020. Two study sites enrolled a total of 24 subjects in the study. Of the 24 subjects enrolled 15 were deemed eligible to undergo surgical implantation and 14 completed the study. All enrolled subjects provided informed consent.
Pre-assignment Details: Per protocol, a subject is considered enrolled upon giving written informed consent. After undergoing the ICF process, subjects completed audiometric testing and speech perception testing to determine eligibility to undergo surgical implantation. Subjects that did not meet the audiometric threshold hearing or speech testing inclusion criteria were discontinued at baseline.
Period: Overall Study
Arm/Group | HiResolution Bionic Cochlear Implant
Started | 24
Completed | 14
Not Completed | 10
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Subject screen failed | 4
Not completed — Surgery denied by subject's insurance carrier | 2

BASELINE CHARACTERISTICS:
Population: Subjects determined eligible for implantation were implanted ear had severe to profound sensorineural hearing (SNHL) loss (PTA > 70 dB HL for 500, 1000, 2000, and 4000 Hz) where SNHL duration was > 3 months and ≤10 year. A moderate SNHL of < 70 dB HL PTA at 500, 1000, 2000, and 4000 Hz was also present in the contralateral (non-implanted) ear. The Consonant-Nucleus-Consonant Word (CNC) word recognition score for both ears was 30% (tested in subject's everyday listening condition for that ear).
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Audiometric Threshold Testing [Mean (Standard Deviation); unit: dB HL]
  Pre-Implant PTA (Ear to be implanted) | 92.1 (21.1)
  Pre-Implant PTA (Contralateral Ear) | 26.0 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Consonant Nucleus-Consonant (CNC) Word Recognition Test (Implanted Ear Only)
Description: The post-implant CNC word scores were compared to preimplant word scores. The CNC monosyllabic word test is a validated test of open-set word recognition ability. The test was administered in quiet at 60 target 0° azimuth) and scored as total number of words correct which is expressed for results/reporting as percentage correct. The CNC word test was the primary speech perception metric used for study inclusion determination and postoperative outcome comparison at defined intervals for this feasibility study. A higher percentage of recognized words represents better hearing of spoken words. The intent is to understand the benefit of the implant treatment option and restoration of auditory input results in improved speech understanding.
Time Frame: Baseline and Twelve months
Population: The primary outcome measure used in this clinical feasibility study was monosyllabic word recognition with the ear to be implanted in quiet using the CNC word test. Subjects that achieved a CNC word recognition score ≤ 30% in the implanted ear and >30% in the contralateral ear. Subjects are tested using their everyday listening condition for each ear.
Measure: Mean (Standard Deviation); unit: percentage of recognized words
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 15
percentage of recognized words
  Baseline CNC Score | 2.13 (7.453)
  12 Month Post Implant CNC score: number analyzed (Participants) | 14
  12 Month Post Implant CNC score | 61.14 (20.240)

2. Primary Outcome: Change in Unaided Hearing Thresholds (Contralateral, Non-Implanted Ear, Only)
Description: Unaided audiometric thresholds compared to preimplant. Standard audiometric procedures were used for the testing of inter-octave frequencies as necessary.
  • Unaided air conduction thresholds using insert earphones at octave frequencies were measured for the contralateral, non-implanted ear at 250, 500, 1000, 2000, 4000 and 8000 Hz. Clinical masking was completed as appropriate.
Time Frame: Baseline and Twelve months
Population: Standard audiometric procedures were used for the testing of inter-octave frequencies as necessary.
  • Unaided air conduction thresholds using insert earphones at octave frequencies were measured for non-implanted ear at 250, 500, 1000, 2000, 4000 and 8000 Hz. Clinical masking was completed as appropriate.
Measure: Mean (Standard Deviation); unit: change in decibels (db)
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 14
change in decibels (db)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at Baseline 250 HZ | 17.14 (7.774)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at 12 Month 250 HZ | 17.14 (8.254)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at Baseline 500 HZ | 17.86 (14.769)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at 12 Month 500 HZ | 20.00 (14.005)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at Baseline 1000 HZ | 23.21 (17.277)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at 12 Month 1000 HZ | 25.71 (18.172)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at Baseline 2000 HZ | 28.57 (21.342)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at the 12 Month 2000 HZ | 28.93 (20.679)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at Baseline 4000 HZ | 35.00 (29.483)
  Pooled Air Conduction Threshold Data for the Contralateral Earat the 12 Month 4000 HZ | 37.86 (31.483)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at Baseline 8000 HZ | 34.29 (31.736)
  Pooled Air Conduction Threshold Data for the Contralateral Ear at 12 Month 8000 HZ | 40.36 (38.203)

3. Primary Outcome: Change in Speech Perception (Bilateral Listening Condition) - Speech Front, Noise Front
Description: AzBio speech scores in speech front, noise front twelve months post implantation compared to preimplant bilateral sentence scores. The AzBio speech testing was the primary speech perception metric used for baseline and postoperative outcome comparison at defined intervals for this feasibility study. A higher percentage of recognized words represents better hearing of spoken words.
Time Frame: Baseline and Twelve months
Population: Speech recognition in noise was measured with the AZBio speech perception test presented in a background of noise in which the target remained at 0° and noise was presented from 0° (speech front).
Measure: Mean (Standard Deviation); unit: percentage of recognized words
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 15
percentage of recognized words
  Baseline Pooled AzBio in Noise Data - Speech Front / Noise Front | 87.39 (15.382)
  Month 12 Pooled AzBio in Noise Data - Speech Front / Noise Front: number analyzed (Participants) | 14
  Month 12 Pooled AzBio in Noise Data - Speech Front / Noise Front | 91.20 (13.08)

4. Primary Outcome: Change in Lateralization Ability Testing (Bilateral Listening Condition)
Description: Lateralization is ability to recognize the location of sound origin compared to preimplantation. The subject was asked to identify if the sentence was heard from the right or left loudspeaker. Scoring was based on the number of sentence locations correctly identified and expressed as a percent average. A higher percent average indicates a better ability to identify sound location.
Time Frame: Baseline and Twelve months
Population: Lateralization ability was measured as the ability to identify the location of a sound presented from a loudspeaker placed at +/- 45° in front of the subject. Test is performed using the participant's bilateral, everyday listening condition using both ears and reported for all subjects at baseline compared to month12.
Measure: Mean (Standard Deviation); unit: percentage of sentences localized
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 15
percentage of sentences localized
  Baseline Pooled Lateralization Ability Data | 72 (21.634)
  Month 12 Pooled Lateralization Ability Data: number analyzed (Participants) | 13
  Month 12 Pooled Lateralization Ability Data | 89.10 (19.522)

5. Primary Outcome: Change in Speech Perception (Bilateral Listening Condition) - Speech Front/Noise to Implanted Ear
Description: AzBio word scores in speech front, noise to implanted ear twelve months post implantation compared to preimplant bilateral sentence scores. The AzBio speech testing was a speech perception metric used for baseline and postoperative outcome comparison at defined intervals for this feasibility study. A higher percentage of recognized words represents better hearing of spoken words.
Time Frame: Baseline to Twelve Months
Population: Speech recognition in noise was measured with the AZBio Speech test presented with the participant at 0° and noise was presented at either 90° or 270° dependent on the implanted ear side.
Measure: Mean (Standard Deviation); unit: percentage of recognized words
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 15
percentage of recognized words
  Baseline Pooled AzBio in Noise Data - Speech Front / Noise to Implanted Ear | 92.15 (15.689)
  Month 12 Pooled AzBio in Noise Data - Speech Front / Noise to Implanted Ear: number analyzed (Participants) | 13
  Month 12 Pooled AzBio in Noise Data - Speech Front / Noise to Implanted Ear | 93.01 (10.165)

6. Primary Outcome: Bilateral Listening Condition (Both Ears - Everyday Listening Condition for Each Ear) - Speech Front /Noise to Non-Implanted Ear.
Description: AzBio speech scores in speech front, noise to the contralateral ear at 12 months post implantation compared to preimplant bilateral sentence scores. The baseline speech perception testing was a speech perception metric used for baseline and postoperative outcome comparison at defined intervals for this feasibility study. A higher percentage of recognized words represents better hearing of spoken words.
Time Frame: Baseline to Twelve Months
Population: Speech recognition in noise was measured with the AZBio Speech test presented with the participant at 0° and noise was presented from either 90° or 270° dependent on the contralateral ear side. Higher percentages score represents a better ability to identify speech source location.
Measure: Mean (Standard Deviation); unit: percentage of recognized words
Arm/Group | HiResolution Bionic Cochlear Implant
Number analyzed (Participants) | 15
percentage of recognized words
  Baseline Pooled AzBio in Noise Data - Speech Front / Noise to Contralateral Ear | 82.24 (19.318)
  Month 12 Pooled AzBio in Noise Data - Speech Front / Noise to Contralateral Ear: number analyzed (Participants) | 13
  Month 12 Pooled AzBio in Noise Data - Speech Front / Noise to Contralateral Ear | 89.10 (19.522)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were recorded and tracked between completion of the informed consent form (signed and dated) and two weeks after the participant's last study visit (approximately 13 months).
Description: All adverse events were reported per subject and classified based on type and frequency. Information recorded included onset date, if the AE was serious, categorization, description, course of action taken, status, and relationship to study device or procedure.
Arm/Group | HiResolution Bionic Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HiResolution Bionic Cochlear Implant (N=15)
Complication at implant site (Surgical and medical procedures) | 1 (1) — Implanted ear
Mild Tinnitus, intermittent - Left Ear (Ear and labyrinth disorders) | 1 (1) — Non-implanted Ear
Moderate Tinnitus, continuous - Right Ear (Ear and labyrinth disorders) | 2 (3) — Implanted Ear
Allergy induced asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Systemic Adverse Events only
Anxiety (General disorders) | 1 (1) — Systemic Adverse Events only
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) — Both implanted and non-implanted ear
Granuloma (General disorders) | 1 (1) — Systemic Adverse Events only
Headache (General disorders) | 1 (1) — Systemic Adverse Events only
Imbalance (General disorders) | 1 (1) — Systemic Adverse Events only
Itching in implanted ear (Ear and labyrinth disorders) | 1 (1) — Implanted ear
Lightheadedness (General disorders) | 1 (1) — Systemic Adverse Events only
Mild ear pressure (Ear and labyrinth disorders) | 1 (1) — Implanted ear
mild head & neck pain post-surgery (General disorders) | 1 (1) — Systemic Adverse Events only
Numbness, discomfort, or pain at or around the pinna (Ear and labyrinth disorders) | 4 (4) — Implanted ear
Pain and Anxiety when wearing external device (General disorders) | 1 (1) — Implanted Ear
Residual hearing loss with a PTA greater than 30dB (Ear and labyrinth disorders) | 9 (9) — Implanted Ear
Sinus Infection (Infections and infestations) | 1 (1) — Systemic Adverse Events only
Small scab superior pole of incision line related to the patient's haircut (General disorders) | 1 (1) — Systemic Adverse Events only
Jaw Pain when chewing (General disorders) | 1 (1) — Systemic Adverse Events only
Soreness, Tenderness, or Pain at or around the incision site (General disorders) | 4 (4) — Implanted ear
Tongue Numbness (General disorders) | 1 (1) — Systemic Adverse Events only
Transient Pain (General disorders) | 1 (1) — Systemic Adverse Events only
Unsteady Gait (General disorders) | 1 (1) — Systemic Adverse Events only
Severe Tinnitus - Left Ear (Ear and labyrinth disorders) | 2 (2) — Implanted ear
Severe Tinnitus - Right ear (Ear and labyrinth disorders) | 2 (2) — Implanted ear
Taste Disturbance (General disorders) | 4 (4)
Vertigo or Dizziness (General disorders) | 7 (7) — Systemic Adverse Events only
Moderate Tinnitus, continuous - Left Ear (Ear and labyrinth disorders) | 1 (1) — Implanted ear
Aural fullness (Ear and labyrinth disorders) | 1 (1) — Implanted ear and Non-implanted Ear

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to submit any publication to Sponsor at least 30 days before submission. Within 30 days, Sponsor advises PI in writing of any information contained therein which is Confidential Information (other than Study Data) or which may impair availability of patent protection for Inventions.

Sponsor has the right to require PI to remove specifically identified CI and/or to delay the publication for an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT02811549/Prot_SAP_000.pdf